CLINICAL TRIAL: NCT00535769
Title: Evaluation of Adherence to Topical Agents: Applying Communication Technology to Improve Sunscreen Use
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Alexandra Kimball, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2007-P-001456
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Skin Cancer
Keywords: topical; medication adherence; adherence; compliance; medication compliance; sunscreen; reminder
MeSH Terms: conditions — Skin Neoplasms; Medication Adherence; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic monitor + no text message (Placebo Comparator): The control or placebo comparator group of subjects will receive the study sunscreen with the attached electronic monitor. They will be instructed to apply sunscreen once a day in the morning to the sun-exposed areas of the body. If the subjects are to have continuous sun exposure (for example, at a beach), they are to re-apply the sunscreen every 3 hours.
  Interventions: Device: Electronic + no text message
- Electronic monitor + Text message (Experimental): The text message experimental group of subjects will receive the study sunscreen with the attached electronic monitor. In addition, this group will receive daily text messages on their cellular phone to remind them to apply the sunscreen. The text message will also contain the daily weather information. This group will also be instructed to apply sunscreen once a day in the morning to the sun-exposed areas of the body. If subjects are to have continuous sun exposure (for example, at a beach), they are to re-apply the sunscreen every 3 hours.
  Interventions: Device: Electronic monitor + text messages

INTERVENTIONS:
Device: Electronic + no text message — Electronic monitor is attached but no text-messages are sent through cellular phones
  Other Names: Electronic monitor without text messages
  Arms: Electronic monitor + no text message
Device: Electronic monitor + text messages — Electronic monitor is attached and text messages are sent through cellphone to remind sunscreen use
  Other Names: Electronic monitor with text message
  Arms: Electronic monitor + Text message

SUMMARY:
The purpose of this study is to determine if using an electronic reminder improves adherence to sunscreen use. The specific study aims are as follows:

1. To determine whether the use of electronic reminder system increases adherence to topical agents.
2. To assess technological feasibility of measuring adherence to topical agents using electronic monitors specially designed for tubes.
3. To assess technological feasibility of providing electronic reminders using cellular phone text-messaging system.
4. To obtain subjects' feedback on the adherence monitoring and reminder system.

DETAILED DESCRIPTION:
We propose to use communication technology to develop a novel means of monitoring and improving adherence to topical agents. We will conduct a randomized, single-blinded, controlled trial to assess the impact of automated reminder system on adherence rates to sunscreens. This study will involve designing an electronic monitoring device specifically for topical agents and creating a platform for an automated reminder system. The electronic monitoring devices will be adaptable to tubes of varying shapes and sizes, and they will send SMS messages to a central server in real-time each time the tube is opened. We will create a text-message reminder system to send reminders to users' cellular phones over a secured network. Our hypothesis is that the electronic monitoring and reminder system will increase patients' adherence to topical agents. We will measure the impact of the intervention on adherence rates and assess patients' views on the reminder system. This project will allow us to engineer a novel device to electronically monitor adherence to topical agents and to use communication technology to change patients' behavior.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of consent, may be men or women.
* Capable of giving informed consent
* Have a cellular phone capable of receiving text messages.
* Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Non-English speaking individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexa B Kimball, MD MPH, Principal Investigator — Brigham and Women's Hospital and Massachusetts General Hospital; April W Armstrong, MD, Study Director — Brigham and Women's Hospital and Massachusetts General Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Armstrong AW, Watson AJ, Makredes M, Frangos JE, Kimball AB, Kvedar JC. Text-message reminders to improve sunscreen use: a randomized, controlled trial using electronic monitoring. Arch Dermatol. 2009 Nov;145(11):1230-6. doi: 10.1001/archdermatol.2009.269. PMID 19917951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: participants must be >18 yo, own a cellular telephone with text-message features, and know how to retrieve text messages.
Groups:
- Control: Electronic Monitor+ no Text Message: The control group of subjects will receive the study sunscreen with the attached electronic monitor. They will be instructed to apply sunscreen once a day in the morning to the sun-exposed areas of the body. If the subjects are to have continuous sun exposure (for example, at a beach), they are to re-apply the sunscreen every 3 hours.
- Electronic Monitor + Text Message: The text message group of subjects will receive the study sunscreen with the attached electronic monitor. In addition, this group will receive daily text messages on their cellular phone to remind them to apply the sunscreen. The text message will also contain the daily weather information. This group will also be instructed to apply sunscreen once a day in the morning to the sun-exposed areas of the body. If subjects are to have continuous sun exposure (for example, at a beach), they are to re-apply the sunscreen every 3 hours.
Period: Overall Study
Arm/Group | Control: Electronic Monitor+ no Text Message | Electronic Monitor + Text Message
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control: Electronic Monitor+ no Text Message | Electronic Monitor + Text Message | Total
Number analyzed (Participants) | 35 | 35 | 70
Age Continuous [Mean (Standard Deviation); unit: years] | 34.3 (14.2) | 32.9 (13.4) | 33.6 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 10 | 11 | 21
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Days the Subjects Are Adherent to Using Sunscreen
Description: Participants' adherence was captured in real time using transmitting electronic monitors. At the end of the 6 week trial, the mean number of days the subjects are adherent to using sunscreen were compared.
Time Frame: 6 weeks
Population: All participants were analyzed
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Control: Electronic Monitor+ no Text Message | Electronic Monitor + Text Message
Number analyzed (Participants) | 35 | 35
days | 12.6 [9.7 to 15.5] | 23.6 [20.2 to 26.9]

2. Secondary Outcome: Usefulness of Text Messaging System
Description: Patients with the text message reminder system were asked their opinion on their satisfaction/ improved adherence to sunscreen application with the use of the messaging system on a scale of 0 to 10 (0, not useful at all; 10,most useful)
Time Frame: 6 weeks
Population: Patients with text messaging system included in analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Usefulness of Text Messaging System: Patients with text reminder system were asked their opinion of the usefulness of message reminder from 0-10 (0, not useful at all; 10,most useful)
Arm/Group | Usefulness of Text Messaging System
Number analyzed (Participants) | 35
units on a scale | 8.31 (1.99)

3. Secondary Outcome: Recalled Frequency of Sunscreen Application
Description: The participants were asked to recall their frequency of sunscreen application based on a 5 point scale (0 never used sunscreen,; 1 forgot to apply 3x weekly,; 2 forgot to apply 1-2x weekly; 3 forgot to apply 1-2x per month; 4 always remembered)
Time Frame: 6 weeks
Population: All participants were assessed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control: Electronic Monitor+ no Text Message | Electronic Monitor + Text Message
Number analyzed (Participants) | 35 | 35
units on a scale | 2.14 (1.17) | 2.42 (0.95)

ADVERSE EVENTS:
Arm/Group | Control: Electronic Monitor+ no Text Message | Electronic Monitor + Text Message
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No